CLINICAL TRIAL: NCT02205567
Title: The Effect of Bergamot on Plasma Lipids, Lipoproteins and Carotid Intima-media Thickness
Brief Title: Bergamot and Cardio-Metabolic Risk Factors
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Manfredi Rizzo, Assistant Professor, University of Palermo
Other Study IDs: BMT14
Record Dates: First submitted 2014-07-29; First posted 2014-07-31 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 2: 1000 mg/day of Bergamot-derived product
  Interventions: Dietary Supplement: Bergamot-derived product
- Group 1: 500 mg/day of Bergamot-derived product
  Interventions: Dietary Supplement: Bergamot-derived product

INTERVENTIONS:
Dietary Supplement: Bergamot-derived product — Group 1: 500mg/day Group 2: 1000mg/day

SUMMARY:
Bergamot-derived products have shown significant effects on plasma lipids. We aim in the present study to evaluate the effect of bergamot on several cardio-metabolic risk markers.

DETAILED DESCRIPTION:
The research hypothesis is to assess whether bergamot reduces plasma lipids (total cholesterol, triglycerides, low-density lipoprotein (LDL)-cholesterol and high-density lipoprotein (HDL)-cholesterol), atherogenic lipoproteins, carotid intima-media thickness (IMT) and liver steatosis in patients with dyslipidemia.

The primary objective is to assess whether bergamot reduces plasma lipids and atherogenic lipoproteins in patients with dyslipidemia.

Primary endpoint: Reduction in plasma lipids and atherogenic lipoproteins. The secondary objective is to assess whether bergamot reduces carotid intima-media thickness (IMT) and liver steatosis in patients with dyslipidemia.

Secondary endpoint: Reduction in IMT and and liver steatosis.

Clinical diagnostic tools will include the measurement of:

1. cIMT, that will be assessed by B-mode real-time ultrasound using a single sonographer (Medison SonoAce Pico, with a probe of 7.5-10.0 MHz) in a standardized manner with fixed angles of insonation;
2. liver steatosis, that will be assessed by by abdominal ultrasound.

Biochemical analyses will include the analysis of:

1. Routine testing of plasma lipids;
2. Atherogenic lipoproteins, e.g. the analysis of 11 distinct lipoproteins including very-low-density lipoprotein (VLDL), 3 intermediate density lipoprotein (IDL) subclasses and 7 low density lipoprotein (LDL) subclasses.

ELIGIBILITY:
Inclusion Criteria:

* elevated LDL-cholesterolemia

Exclusion Criteria:

* severe hepatic or renal diseases

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult subjects with dyslipidemia
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in plasma lipids | baseline and 6 months
  We will measure at baseline and after 6 months the following plasma lipids concentrations: total cholesterol, triglycerides, LDL-cholesterol and HDL-cholesterol.

SECONDARY OUTCOMES:
Change from baseline in atherogenic lipoproteins, carotid intima-media thickness (IMT) and liver steatosis | baseline and 6 months
  We will measure at baseline and after 6 months carotid IMT by color doppler ultrasound, atherogenic lipoproteins by electrophoresis and liver steatosis by abdominal ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Montalto, MD, Study Director — University of Palermo, Italy
Locations (1):
- University Hospital of Palermo, Palermo, PA, Italy